CLINICAL TRIAL: NCT07332091
Title: A Phase 2, Multicenter, Randomized, Placebo-controlled, Double-blind Study of the Efficacy and Safety of Vamifeport in Adult Subjects With HFE-related Hereditary Hemochromatosis (FERROCLEAR Study)
Brief Title: Efficacy and Safety of Vamifeport in Adult Participants With Homeostatic Iron Regulator Gene (HFE)-Related Hereditary Hemochromatosis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CSL624_2001; 2025-523793-16-00 (Other: EU CT Number)
Record Dates: First submitted 2026-01-08; First posted 2026-01-12 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Homeostatic Iron Regulator Gene-related Hereditary Hemochromatosis
Keywords: Small Molecule Ferroportin Inhibitor; Hereditary hemochromatosis; Iron overload
MeSH Terms: conditions — Hemochromatosis; Iron Overload

STUDY DESIGN:
Intervention Model Description: This is multicenter, randomized, placebo-controlled double-blind, parallel-group study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Vamifeport Low Dose (Experimental): Participants will receive a low dose of vamifeport orally, twice daily (BID) up to Day 360.
  Interventions: Drug: Vamifeport
- Vamifeport High Dose (Experimental): Participants will receive a high dose of vamifeport orally, BID up to Day 360.
  Interventions: Drug: Vamifeport
- Placebo (Placebo Comparator): Participants will receive placebo matching vamifeport low and high doses orally, BID up to Day 360.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vamifeport — Vamifeport capsule administered orally.
  Arms: Vamifeport High Dose; Vamifeport Low Dose
Drug: Placebo — Placebo capsule matching IP administered orally.
  Arms: Placebo

SUMMARY:
This is a phase 2, multicenter, randomized, placebo-controlled, double-blind, parallel-group, proof-of-concept study to assess vamifeport in adult participants with homeostatic iron regulator gene-related hereditary hemochromatosis (HFE-HH). The primary objective of the study is to assess the effect of vamifeport treatment on magnetic resonance imaging (MRI)-based liver iron concentration (LIC) in adult participants with HFE-HH.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥ 18 years) and has provided written informed consent.
* Confirmed diagnosis of HFE-HH in medical history.
* Evidence of iron overload as shown by:

  * TSAT > 45% (confirmed at 2 visits, at least 14 days apart) at Screening; and
  * Serum ferritin ≥ 200 nanogram per milliliter (ng/mL) and < 5000 ng/mL (confirmed at 2 visits, at least 14 days apart) at Screening; and
  * MRI-based LIC between 3 and 16 mg/g (53.7 and 286.5 millimol per kilogram [mmol/kg]) dry weight (dw) at Screening.
* Body mass index between 18.5 and 32 kilograms per meter squared (kg/m^2).

Exclusion Criteria:

* Clinically relevant laboratory abnormalities, 12-lead electrocardiogram (ECG) findings, or medical history.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2026-02-08 (Estimated); Primary Completion 2028-03-06 (Estimated); Study Completion 2028-04-06 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in magnetic resonance imaging (MRI)-based liver iron concentration (LIC) | At Baseline and Day 360

SECONDARY OUTCOMES:
Number of participants with treatment-emergent adverse events (TEAEs) | Up to Day 390
Percentage of participants with TEAEs | Up to Day 390
Number of participants with treatment-emergent serious adverse events (SAEs) | Up to Day 390
Percentage of participants with treatment-emergent SAEs | Up to Day 390
Number of participants with clinically significant change from baseline in clinical safety laboratory tests and 12-lead electrocardiogram (ECG) | From Baseline to Day 390
  Clinical safety laboratory tests will include hematology, biochemistry and coagulation.
Percentage of participants with clinically significant change from baseline in clinical safety laboratory tests and 12-lead ECG | From Baseline to Day 390
  Clinical safety laboratory tests will include hematology, biochemistry and coagulation.
Change from baseline in transferrin saturation (TSAT) (measured at trough) | From Baseline to Day 360
Number of participants with TSAT less than or equal to (<=) 45% (measured at trough) | From Baseline to Day 360
Percentage of participants with TSAT <= 45% (measured at trough) | From Baseline to Day 360
Number of participants with 25% reduction in MRI-based LIC | At Day 180 and 360
Number of participants with 50% reduction in MRI-based LIC | At Day 180 and Day 360
Number of participants with TSAT ≤ 45% or MRI-based LIC < 5 milligrams per gram (mg/g) | At Day 360
Number of participants with TSAT ≤ 45% or MRI-based LIC < 2 mg/g | At Day 360
Change from baseline in joint pain score in a visual analog scale (VAS) | From Baseline to Day 360
  The VAS is a single-item questionnaire. Participants will be asked to record their joint pain at its worst over the previous week, from 0 (No pain) to 10 (Worst possible pain).
Change from baseline in modified fatigue impact scale (MFIS) total score | From Baseline to Day 360
  Participants will be asked to read a list of 21 statements and assess how often fatigue has affected them in terms of physical, cognitive, and psychosocial functioning, over the previous 4 weeks, using a 5-point scale from 0 (Never) to 4 (Almost always). The total score is obtained by summing the scores of all the 21 items. Higher scores indicate a greater impact of fatigue on a participant's activities.
Change from baseline in health-related quality of life: EuroQoL 5-dimension 5-level instrument (EQ-5D-5L) | From Baseline to Days 180, 360, and 390
  The EQ-5D-5L is a standardized measure of health status that provides a simple, generic measure of health for clinical and economic appraisal. Participants will complete the questionnaire based on their health on that day. The EQ-5D-5L descriptive profile includes 5 dimensions: mobility, self-care, usual activities, pain / discomfort, and anxiety / depression. Participants will rate each dimension based on 5 levels of severity: no problems, slight problems, moderate problems, severe problems, and extreme problems. A higher score indicates a more severe outcome than a lower score.
Change from baseline in health-related quality of life: VAS (Arthralgia) | From Baseline to Day 180, 360, and 390
  The VAS is a single-item questionnaire. Participants will be asked to record their joint pain at its worst over the previous week, from 0 (No pain) to 10 (Worst possible pain).
Change from baseline in health-related quality of life: Patient global impression of change in clinical status | From Baseline to Day 180, 360, and 390
  The PGI - Change (PGI-C) instrument is a self-reported measure that reflects belief about the efficacy of treatment. Participants will be asked to rate the change in their overall symptoms since they started taking investigational product (IP) on a 5-point scale, ranging from 1 (Much improved) to 5 (Much worse). A lower score reflects an improvement in clinical status.
Change from baseline in health-related quality of life: Patient global impression of severity | From Baseline to Day 180, 360, and 390
  The PGI - Severity (PGI-S) instrument is a self-reported questionnaire and consists of 1 item that measures disease severity. Participants will be asked to rate the severity of their overall symptoms over the previous week on a 5-point scale from 1 (None) to 5 (Very severe). A higher score reflects a more severe outcome than a lower score.
Change from baseline in health-related quality of life: MFIS physical, cognitive, and psychosocial subscales | From Baseline to Day 180, 360, and 390
  Participants will be asked to read a list of 21 statements and assess how often fatigue has affected them in terms of physical, cognitive, and psychosocial functioning, over the previous 4 weeks, using a 5-point scale from 0 (Never) to 4 (Almost always).
  Items on the MFIS will be aggregated into 3 subscales (Physical, Cognitive, or Psychosocial). Higher scores indicate a greater impact of fatigue on a participant's activities.
Vamifeport plasma concentrations after a single dose | At Day 1
Vamifeport plasma concentrations at steady state | At Days 15, 180, and 360
Change from baseline in total serum iron (measured at trough) | From Baseline to Day 360
Change from baseline in serum ferritin (measured at trough) | From Baseline to Day 360
Frequency of rescue therapy use | Up to Day 390
  For assessment of this outcome measure, data will be collected retrospectively from 1 year before baseline as well as during the study (up to Day 390).
Duration of rescue therapy use | Up to Day 390
  For assessment of this outcome measure, data will be collected retrospectively from 1 year before baseline as well as during the study (up to Day 390).
Time to first use of rescue therapy | Up to Day 360

CONTACTS AND LOCATIONS:
Locations (96):
- United States (18):
  - Banner MD Anderson, Gilbert, Arizona
  - Infinity Clinical Trials, San Diego, California
  - Medical Oncology Associates of San Diego, San Diego, California
  - Green Leaf Clinical Trials, Jacksonville, Florida
  - Indiana University Health University Hospital, Indianapolis, Indiana
  - Ochsner Medical Complex - High Grove, Baton Rouge, Louisiana
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - American Oncology Partners, PA dba The Center for Cancer and Blood Disorders, Bethesda, Maryland
  - James M. Stockman Cancer Institute, Frederick, Maryland
  - University of Michigan Health System (UMHS), Ann Arbor, Michigan
  - Aspirus St. Luke's Clinic - Duluth - Oncology & Hematology, Duluth, Minnesota
  - Hunterdon Hematology Oncology, LLC, Flemington, New Jersey
  - Derald H. Ruttenberg Treatment Center, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke University Medical Center (Duke South Clinics) -40 Duke Medicine Cir, Durham, North Carolina
  - Hightower Clinical - Oklahoma Cancer Center, Oklahoma City, Oklahoma
  - Intermountain Medical Center, Murray, Utah
  - Washington State Univ Elson S. Floyd College of Medicine, Spokane, Washington
- Australia (5):
  - Royal Brisbane and Women's Hospital, Brisbane
  - Gallipoli Medical Research, Chandler
  - Monash Medical Centre, Clayton
  - Trials West, Perth
  - Westmead Hospital, Westmead
- Austria (3):
  - Medical University of Innsbruck, Innsbruck
  - Ordensklinikum Linz - Barmherzige Schwestern, Linz
  - Medical University Vienna, Vienna
- Belgium (5):
  - Universitair Ziekenhuis Antwerpen (UZA), Edegem
  - Ghent University Hospital, Ghent
  - UZ Brussel, Jette
  - Centre Hospitalier Universitaire de Liège (CHU de Liège), Liège
  - CHU UCL Namur - Site Godinne, Yvoir
- Canada (3):
  - Libin Cardiovascular Institute University of Calgary, Calgary
  - St. Josephs Healthcare Hamilton, Hamilton
  - University of Manitoba, Winnipeg
- Czechia (3):
  - Fakultní Nemocnice Brno, Brno
  - Fakultni nemocnice Ostrava, Ostrava
  - Institut Klinicke a Experimentalni Mediciny, Prague
- Denmark (3):
  - Aarhus University Hospital, Aarhus
  - Bispebjerg Hospital, Copenhagen
  - Copenhagen University Hospital - Hvidovre, Hvidovre
- France (11):
  - Aphp Avicenne, Bobigny
  - Chu Dupuytren, Limoges
  - CRMR Maladies du Globule Rouge, Hôpital de la Timone, Marseille
  - CHU de Montpellier- Hôpital Saint Eloi, Montpellier
  - GHRMSA, Mulhouse
  - CHU de Bordeaux - Hôpital Haut Leveque, Pessac
  - Centre Hospitalier Lyon Sud/Hospices Civils de Lyon, Pierre-Bénite
  - Chu Rennes, Rennes
  - Centre Hospitalier de Saint Brieuc, Saint-Brieuc
  - CHU Toulouse, Toulouse
  - Hôpital Paul Brousse, Villejuif
- Germany (4):
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - University Hospital Heidelberg, Heidelberg
  - EUGASTRO GmbH, Leipzig
  - MVZ für Innere Medizin Weinheim, Weinheim
- Ireland (3):
  - Cork University Hospital, Cork
  - Beaumont Hospital, Dublin
  - Connolly Hospital Blanchardstown, Dublin
- Italy (6):
  - ASL Brindisi - Presidio Ospedaliero Di Summa - Perrino, Brindisi
  - Fondazione IRCCS Ca Granda Ospedale Maggiore Policlinico, Milan
  - University Hospital of Modena, Modena
  - Fondazione IRCCS San Gerardo dei Tintori, Monza
  - AORN Cardarelli, Naples
  - University of Verona - Azienda Ospedaliera Universitaria Integrata Verona, Verona
- Netherlands (3):
  - Auckland City Hospital, Auckland
  - Maastricht UMC, Maastricht
  - Radboud UMC, Nijmegen
- Poland (3):
  - Instytut Hematologii i Transfuzjologii, Warsaw
  - Specjalistyczny Szpital im. Alfreda Sokolowskiego, Wałbrzych
  - Wojewodzki Szpital im. J Gromkowskiego we Wroclawiu, Wroclaw
- Romania (5):
  - Spitalul Clinic de Urgenta Prof Dr Agrippa Ionescu-Balotesti, Baloteşti
  - Bistrița County Emergency Clinical Hospital, Bistriţa
  - Coltea Clinical Hospital, Bucharest
  - L'Institute Oncologique Prof. Dr. Ion Chiricuta (IOCN), Cluj-Napoca
  - Prof. Dr.Octavian Fodor Regional Institute of Gastroenterology-Hepatology, Cluj-Napoca
- Spain (7):
  - Hospital Universitari Germans Trias i Pujol, Badalona
  - Hospital Clinic Barcelona, Barcelona
  - HUGC Doctor Negrin, LAS Palmas de GC
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Puerta de Hierro - Majadahonda, Majadahonda
  - Althaia Foundation. Hospital Sant Joan de Deu de Manresa, Manresa
  - Hospital Universitario Virgen del Rocío, Seville
- Switzerland (3):
  - University Hospital Inselspital Bern, Bern
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - Epatocentro Ticino, Lugano
- United Kingdom (11):
  - Royal Victoria Hospital, Belfast
  - University Hospitals Bristol and Weston NHS trust, Bristol Haematology and Oncology Centre, Bristol
  - Royal Liverpool University Hospital, Liverpool
  - King's College Hospital, London
  - St Thomas Hospital, London
  - Norfolk and Norwich University Hospital, Norwich
  - Nottingham University Hospitals City Campus, Nottingham
  - John Radcliffe Hospital - Oxford University Hospitals NHS, Oxford
  - Derriford Hospital, Plymouth
  - University Hospital Southampton NHS Foundation Trust, Southampton
  - South Warwickshire University Foundation Trust, Warwick

IPD SHARING:
Plan to Share IPD: Yes
CSL will consider on a case-by-case basis requests to share Individual Patient Data (IPD) with external bona-fide, qualified scientific and medical researchers. For information on the process and requirements for submitting a voluntary data sharing request for IPD, please contact CSL at clinicaltrials@cslbehring.com.
Supporting Information: Study Protocol, SAP
Time Frame: Requests for IPD will generally be considered once review by major regulatory authorities (ie FDA, EMA) is complete and the primary publication is available.
Access Criteria: Proposed research should seek to answer a previously unanswered important medical or scientific question.
  Applicable country specific privacy and other laws and regulations will be considered and may prevent sharing of IPD.
  If the request is approved and the researcher has executed an appropriate data sharing agreement, IPD that has been appropriately anonymized will be available.